CLINICAL TRIAL: NCT00003266
Title: Double-Blind Randomized Trial of Methylphenidate for Alleviation of Fatigue and Lethargy Associated With Interferon Alpha 2b
Brief Title: Methylphenidate in Treating Patients With Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: CDR0000066161; E-2Z96; NCI-P98-0130
Record Dates: First submitted 1999-11-01; First posted 2003-10-28 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Fatigue; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; fatigue
MeSH Terms: conditions — Fatigue | interventions — Methylphenidate

INTERVENTIONS:
Drug: methylphenidate hydrochloride
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Methylphenidate may relieve some of the side effects of chemotherapy in patients with melanoma. It is not known whether receiving methylphenidate is more effective than receiving no further therapy in treating patients with melanoma.

PURPOSE: Randomized phase III trial to determine if methylphenidate is more effective than no further therapy for the relief of fatigue and drowsiness in treating patients with melanoma who have received high-dose interferon alfa for 8-24 weeks.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether methylphenidate decreases fatigue and lethargy in cancer patients receiving interferon alfa. II. Determine whether the use of methylphenidate in this patient population decreases the number of dose reductions of interferon alfa due to toxicities other than myelosuppression or elevated liver function tests. III. Assess whether efficacy or toxicity of methylphenidate in this patient population is concentration dependent. IV. Compare the fatigue subscale and the proposed Brief Fatigue Inventory.

OUTLINE: This is a randomized, double-blind, placebo-controlled, two arm study. Patients are stratified according to initial fatigue level (high vs moderate), and treatment with tumor vaccine (yes vs no). Patients are randomized to one of two treatment arms. Arm I: Patients receive oral methylphenidate twice daily. Arm II: Patients receive oral placebo twice daily. Treatment is continued for 21 consecutive days with dose escalations as tolerated and as needed by patient judgement, followed by an additional week to evaluate the effect of drug withdrawal. Patients are contacted by telephone at least twice weekly during the 21 day treatment and 7 day washout phase to assess adverse or rebound effects. Before the study begins and at weekly clinic visits for the 4 week study period, patients complete a series of questionnaires to measure mood, levels of fatigue and lethargy, and sense of well being. Patients also keep a short daily diary of study medication doses and degree of tiredness. Patients are followed every 3 months for 2 years, then every 6 months for the next 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 200 patients will be accrued into this study within 39 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: On interferon alfa-2b treatment for at least 8 weeks Dose must be stable for 2 weeks prior to and during study Fatigue level at least 4 on the Symptom and Fatigue Self Evaluation Form (0 none, 10 worst possible)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Not specified Life expectancy: More than 4 weeks Hematopoietic: Hematocrit at least 30% Hepatic: Not specified Renal: Creatinine no greater than 2.0 mg/dL Other: No history of any of the following: Chronic use of anticonvulsants Seizure disorder Motor tics Glaucoma Family history or diagnosis of Tourette's disorder No allergic reaction or hypersensitivity to methylphenidate Cognitively able to participate Not incarcerated Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: See Disease Characteristics No monoamine oxidase inhibitors within 2 months

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 1999-10-12 (Actual); Primary Completion 2002-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul R. Hutson, PharmD, Study Chair — University of Wisconsin, Madison
Locations (59):
- United States (57):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Stanford University Medical Center, Stanford, California
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - Veterans Affairs Medical Center - Gainsville, Gainesville, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - CCOP - Ochsner, New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - New England Medical Center Hospital, Boston, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Veterans Affairs Medical Center - New York, New York, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - MBCCOP-Our Lady of Mercy Cancer Center, The Bronx, New York
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Ireland Cancer Center, Cleveland, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Veterans Affairs Medical Center - Pittsburgh, Pittsburgh, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - Veterans Affairs Medical Center - Tennessee Valley Healthcare System - Nashville Campus, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
- MBCCOP - San Juan, San Juan, Puerto Rico
- Pretoria Academic Hospitals, Pretoria, South Africa